CLINICAL TRIAL: NCT01602874
Title: Multicenter, Randomized, And Double-Blind Study To Evaluate The Safety Of Tigecycline Versus A Ceftriaxone Regimen In The Treatment Of Complicated Intra-Abdominal Infections And Community-Acquired Pneumonia In Subjects Of 8-17 Years
Brief Title: Study Evaluating Tigecycline Versus Ceftriaxone In Complicated Intra-Abdominal Infections & Community Acquired Pneumonia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3074K4-3340; B1811003
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Community Acquired Bacterial Pneumonia; Complicated Intra-Abdominal Infection
Keywords: children; pediatry; pneumonia; intra-abdominal; infection
MeSH Terms: conditions — Pneumonia; Infections | interventions — Tigecycline; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A. Tigecycline (Experimental)
  Interventions: Drug: Tigecycline
- B. Ceftriaxone regimen (Active Comparator)
  Interventions: Drug: cIAI: Ceftriaxone with metronidazole, plus if applicable aminoglycoside; Drug: CAP: Ceftriaxone, plus if applicable oral clarithromycin

INTERVENTIONS:
Drug: Tigecycline — Subject with cIAI:
  Dosing information for subjects 8 to 11 years old is currently under investigation and will be determined later. Subjects 12 to 17 years old will receive tigecycline 50 mg IV every 12 hours, metronidazole placebo IV will be administered every 8 hours. In addition, at the discretion of the investigator, an aminoglycoside placebo IV may also be administered.
  Other Names: Tygacil
  Arms: A. Tigecycline
Drug: Tigecycline — Subject with CAP:
  IV therapy period: Dosing information for subjects 8 to 11 years old is currently under investigation and will be determined later. Subjects 12 to 17 years old will receive tigecycline 50 mg IV every 12h. At the discretion of the investigator oral clarithromycin placebo may be given every 12h.
  Oral therapy period: If oral switch criteria are met, on or after Day 4 amoxicillin/clavulanate may be prescribed (40 mg/kg per day divided into 3 equal doses, maximum of 500 mg/dose to subjects weighing less than 40 kg and 500 mg every 8h to subjects weighing 40 kg or greater). In addition, if oral clarithromycin or placebo had been given during the IV period, oral clarithromycin may be given every 12h (7.5 mg/kg, maximum dose 500 mg for subjects 8 to 11 years old, 500 mg for subjects 12 to 17 years old).
  Other Names: Tygacil
  Arms: A. Tigecycline
Drug: cIAI: Ceftriaxone with metronidazole, plus if applicable aminoglycoside — Subject with cIAI:
  Subjects will receive ceftriaxone 35 mg/kg (maximum of 1 g/dose) IV every 12 hours, metronidazole 10 mg/kg (maximum of 1 g/dose) IV will be administered every 8 hours.
  In addition, at the discretion of the investigator, an aminoglycoside IV (adjusted dose if necessary) may also be given.
  Arms: B. Ceftriaxone regimen
Drug: CAP: Ceftriaxone, plus if applicable oral clarithromycin — Subject with CAP:
  IV therapy period: Subjects will receive ceftriaxone 35 mg/kg (maximum of 1 g/dose) IV every 12h. At the discretion of the investigator, oral clarithromycin may be given every 12h (7.5 mg/kg, maximum dose 500 mg for subjects 8 to 11 years old, 500 mg for subjects 12 to 17 years old).
  Oral therapy period: If oral switch criteria are met, on or after Day 4 amoxicillin/clavulanate may be prescribed (40 mg/kg per day divided into 3 equal doses, maximum of 500 mg/dose to subjects weighing less than 40 kg and 500 mg every 8h to subjects weighing 40 kg or greater). In addition, if oral clarithromycin or placebo had been given during the IV period, oral clarithromycin may be given every 12h (7.5 mg/kg, maximum dose 500 mg for subjects 8 to 11 years old, 500 mg for subjects 12 to 17 years old).
  Arms: B. Ceftriaxone regimen

SUMMARY:
The main purpose of this study is to compare the safety of tigecycline versus a ceftriaxone regimen in pediatric subjects (aged 8 to 17 years) with complicated intra-abdominal infections (cIAI) and community acquired pneumonia (CAP).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 8 to 17 years old. Children with bone maturation less than 8 years old should be enrolled with caution due to potential risk of tooth discoloration.
* Have a diagnosis of a serious infection (complicated intra-abdominal infections [cIAI] or community acquired pneumonia [CAP] as applicable) requiring hospitalization and administration of IV antibiotic therapy.
* Criteria related indication (cIAI or CAP - as applicable), e.g., sign of systemic infection, signs and symptom.

Exclusion Criteria:

* Subject with any concomitant illness/condition that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in and/or completion of the study, or could preclude the evaluation of the subject's response (e.g., life expectancy <30 days).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy response (cure, failure, or indeterminate) at the test of cure (TOC) visit for 2 co-primary populations: the clinically evaluable (CE) and clinical modified Intent-to-Treat (c-mITT) populations | 2 to 7 weeks for cIAI and 2 to 5 weeks for CAP

SECONDARY OUTCOMES:
Clinical response at the IV last day of therapy (LDOT) for co-primary populations: the CE and c-mITT populations | 5 days to 4 weeks for cIAI and 5 days to 2 weeks for CAP
Clinical response at follow up (FUP) visits for co-primary populations: the CE and c-mITT populations | 5 to 9 weeks for cIAI and 5 to 7 weeks for CAP
Microbiological response at the subject and the pathogen level | 5 to 9 weeks for cIAI and 5 to 7 weeks for CAP
Response rate by pathogen and minimum inhibitory concentration (MIC) value | 5 to 9 weeks for cIAI and 5 to 7 weeks for CAP
Response rates for polymicrobial/monomicrobial infections, and susceptibility evaluations | 5 to 9 weeks for cIAI and 5 to 7 weeks for CAP

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3074K4-3340&StudyName=Study%20Evaluating%20Tigecycline%20Versus%20Ceftriaxone%20In%20Complicated%20Intra-Abdominal%20Infections%20%26%20Community%20Acquired%20Pneumonia